CLINICAL TRIAL: NCT03761836
Title: Program Evaluation and Active Adverse Event Surveillance for Initial Implementation of WHO Prequalified ShangRing™ Circumcision in Mozambique
Brief Title: Evaluation and Adverse Event Surveillance for Initial Implementation of ShangRing Circumcision in Mozambique
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding no longer available
Sponsor: Jhpiego (Other)
Collaborators: Ministry of Health, Mozambique (Other Government); Centers for Disease Control and Prevention (U.S. Federal Agency); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JHSPH IRB 8231
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Circumcision, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ShangRing (Experimental): Males aged 13 years and above will undergo circumcision through ShangRing procedure, with regular follow-up visits to evaluate pain, wound healing and incidence of adverse events. The ShangRing will be removed after 7 days, with a last follow-up visit at 60 days.
  Interventions: Device: ShangRing

INTERVENTIONS:
Device: ShangRing — The ShangRing™ is a device for male circumcision that was invented by Jian Zhong Shang and has been on the Chinese market since 2005. It consists of a sterile device with two concentric medical grade plastic rings: an inner ring with a silicone band and an outer, hinged ring. The inner ring fits inside the outer ring which will lock when snapped together. It currently holds a European Conformity (CE) mark, an EN ISO certificate, and is FDA approved. Clinical data from ShangRing studies in Africa were reviewed by the WHO Technical Advisory Group (TAG) on Innovations in Male Circumcision in January 2013 and were found to meet its clinical requirements. The ShangRing manufacturer was accepted by the WHO Prequalification Programme for Male Circumcision Devices in 2015.

SUMMARY:
This is a single-arm interventional study of 1000 male circumcision procedures using the ShangRing device. The primary objective of the study is to enhance understanding of the potential clinical and operational challenges and opportunities that may be associated with widespread use of ShangRing™ device for circumcision in different settings in Mozambique. Specific objectives are: 1) To monitor the proportion of men who choose circumcision through the WHO-prequalified, FDA-approved ShangRing™ device in routine voluntary medical male circumcision (VMMC) service delivery settings where standard surgical methods of circumcisions are available; and 2) To ensure safety during initial implementation of the ShangRing™ device and confirm that adverse event rates are comparable to those found during implementation in other sub-Saharan countries.

DETAILED DESCRIPTION:
This is a single-arm interventional study of 1000 male circumcision procedures using the ShangRing device. The primary objective of the study is to enhance understanding of the potential clinical and operational challenges and opportunities that may be associated with widespread use of ShangRing™ device for circumcision in different settings in Mozambique. Specific objectives are:

1. To monitor the proportion of men who choose circumcision through the WHO-prequalified, FDA-approved ShangRing™ device in routine voluntary medical male circumcision (VMMC) service delivery settings where standard surgical methods of circumcisions are available; and
2. To ensure safety during initial implementation of the ShangRing™ device and confirm that adverse event rates are comparable to those found during implementation in other sub-Saharan countries.

Population: 1000 males aged 13 years and above who are seeking male circumcision; 3 clinic sites

Duration: Approximately 3 months of recruitment, 60 days follow-up per participant; total duration expected to be approximately 6 months in the field.

Sample size: Cumulative target of 1000 ShangRing™ procedures, based on guidance contained in the WHO Framework for clinical evaluation of devices for male circumcision. The WHO TAG on Innovations in Male Circumcision recommends active follow-up of the first 1000 clients when a new device is introduced into a program or as a new program is implemented.

Data analysis plan: Baseline demographic and behavioral characteristics of ShangRing™ clients will be summarized using counts and percentages. Association between these variables and selected outcome variables (e.g. AEs, failure to return for device removal, preference for Shang Ring) will be examined through cross tabulations and tests of association (e.g. Chi square statistics).

Data quality assurance: Data quality control efforts will include members of the national VMMC Technical Working Group, including local ShangRing™ Trainers of Trainers, conducting scheduled site assessments/monitoring as follows: Prior to the start of the active surveillance (site initiation) using site assessment checklist; and every month using a VMMC quality assessment checklist. There will be regular monthly supervision visits to the facilities to ensure proper record filing and storage of physical forms. Data will be entered into an electronic system by trained data personnel at the facility level. This data will be reviewed actively and regularly through the central database on a periodic basis. The PI, lead local investigator and co-investigators will regularly monitor and evaluate data for completeness and specifically to monitor for any adverse events that may preclude or terminate the study early. The electronic system will be monitored regularly and by limited access of study personnel.

ELIGIBILITY:
Inclusion Criteria:

1. Male, 13 years old and above
2. Agrees to return to the facility where circumcision procedure is done for device removal on day 7 and to have home or off-site visits if deemed necessary by the ShangRing™ providers
3. Is able and willing to provide a valid physical address of residence and at least one alternate address (address of employer, school, or friend/relative) for tracing
4. Is able and willing to provide a valid primary phone number and at least one alternate phone number (phone number of friend/relative) and agrees to be contacted via that alternate number and person. This will facilitate telephone-based follow-up should he not return for the scheduled post-removal follow-up visits.

Exclusion Criteria:

1. Males below 13 years of age
2. Males for whom the correct fitting size of ShangRing™ Device is not available
3. Anatomical abnormalities including adhesions
4. Cognitive impairment
5. Any health condition (reported or observed) that ShangRing™ providers deem a contraindication to the procedure. These may include history of diabetes, peripheral vascular disease, cancer, bleeding disorders, and/or current moderate or severe infectious illness
6. HIV - positive (although may still undergo surgical circumcision)
7. Anatomical variations and anomalies of genitalia
8. Hypospadias, epispadias, or other urethral anomaly
9. Hydrocele
10. Scrotal hernia
11. Other genital anomaly or disease including infectious or traumatic ulcers
12. Dermatitis of the penis or foreskin
13. Genital warts
14. Urethral discharge
15. Balanitis

Min Age: 13 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of ShangRing clients who experience moderate and severe adverse events | 60 days postoperative
  Circumcision-related adverse events are classified as moderate and severe per standardized protocol definitions

SECONDARY OUTCOMES:
Proportion of eligible men who chose ShangRing procedure | Preoperative
  ShangRing will be offered as a neutral alternative to conventional surgery or other available methods
Proportion of ShangRing™ clients who fail to return for device removal on day 7 | 7 days postoperative
  Calculated by site and disaggregated by age group
Pain scores on Visual Analog Scale | Within 48 hours postoperative
  Peri- and post-operative pain scores as determined by visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Necochea, MD, MPH, Principal Investigator — Jhpiego
Locations (3):
- Mozambique (3):
  - Matola II Health Center, Matola, Maputo Province
  - September 17 Health Center, Quelimane, Zambezia Province
  - Infulene Psychiatric Hospital, Maputo

IPD SHARING:
Plan to Share IPD: Undecided